CLINICAL TRIAL: NCT02328794
Title: Randomized Clinical Trial to Reduce Harm From Tobacco
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Vitality Institute (Unknown)
Responsible Party: Principal Investigator, Scott Halpern, Assistant Professor of Medicine, University of Pennsylvania
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 820451
Record Dates: First submitted 2014-12-15; First posted 2014-12-31 (Estimated); Last update posted 2017-05-02 (Actual); Status verified 2017-05

CONDITIONS: Smoking Cessation
Keywords: smoking cessation; behavioral economics; e-cigarettes; NRT
MeSH Terms: conditions — Smoking Cessation; Vaping

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- Control (Active Comparator): Participants randomized to this arm will receive a standardized Vitality program aimed at promoting tobacco cessation. This program includes existing employee benefits for quitting and the use of text/email messages to encourage tobacco cessation. No incentives will be given to participants randomized to this arm. Free cessation aids will not be available to participants in this arm. They will receive compensation for completing study related activities (sample submissions).
  Interventions: Behavioral: Control
- E-cigarette free access (Experimental): Participants randomized to this experimental arm will receive the standardized program including text/email messaging and will have access to free e-cigarettes only. These products can be ordered directly, free of charge, through the web-based interface. No incentives will be given to participants randomized to this arm. They will receive compensation for completing study related activities (sample submissions).
  Interventions: Behavioral: E-cigarette free access
- E-cigarette/NRT/Zyban/Chantix Choice (Experimental): Participants randomized to this experimental arm will receive the standardized program including text/email messaging and will have access to free e-cigarettes, conventional Nicotine Replacement Therapy (NRT), Zyban, or Chantix. Each of these can be ordered directly, free of charge, through the web-based interface. No incentives will be given to participants randomized to this arm. They will receive compensation for completing study related activities (sample submissions).
  Interventions: Behavioral: E-cigarette/NRT/Zyban/Chantix Choice
- Outcome Incentive arm (Experimental): Participants randomized to this experimental arm will receive the standardized program and access to free e-cigarettes, NRT, Zyban, or Chantix. In addition, they will also be able to earn incentives across six months for testing negative for tobacco use (see Incentive payout, below). They will also receive compensation for completing study related activities (sample submissions).
  Interventions: Behavioral: Outcome Incentive arm
- Loss framing incentive arm (Experimental): Participants randomized to this experimental arm will receive the standardized program and access to free e-cigarettes, NRT, Zyban, or Chantix. In addition they will also be able to earnincentives across six months through a pre-funded deposit or precommitment account. They will be notified that money has been placed into an account for them. At each time point they will lose a portion (see below) of this initial funding if they do not provide biochemical evidence of abstinence. They will also receive compensation for completing study related activities (sample submissions).
  Interventions: Behavioral: Loss framing incentive arm

INTERVENTIONS:
Behavioral: E-cigarette free access — Participants in this arn will be given free access to e-cigarettes to help quit smoking
  Arms: E-cigarette free access
Behavioral: E-cigarette/NRT/Zyban/Chantix Choice — Participants in this arn will be given free access to cessation aids to help quit smoking
  Arms: E-cigarette/NRT/Zyban/Chantix Choice
Behavioral: Outcome Incentive arm — Participants in this arm will be earn incentives across 6 months for verified abstinence.
  Arms: Outcome Incentive arm
Behavioral: Loss framing incentive arm — Participants in this arm will be told they have a pre-funded account with money that is theirs if they quit smoking.
  Arms: Loss framing incentive arm
Behavioral: Control — Participants will have access to information and advice on quitting smoking. This is a control and no actual intervention will be applied.
  Arms: Control

SUMMARY:
Using the NIH-funded Way to Health platform, the investigators will conduct this smoking cessation RCT among Vitality/Discovery beneficiaries. The investigators will be able to determine the effectiveness of 4 different interventions aimed at smoking cessation, two of which are incentive structures that are each grounded in behavioral economic principles. The other interventions will determine the effectiveness of various cessation aids, including electronic cigarettes and text messaging, on smoking cessation. This study will be conducted as an opt-out procedure where participants are automatically enrolled in the program but have the choice to unenroll if they so chose. This pragmatic approach will allow us to investigate the effects of such programs in an employee based population that can be easily mimicked in other employee based populations.

DETAILED DESCRIPTION:
Overall objectives Our primary objective is to determine which of four interventions improve smoking cessation rates in beneficiaries of the Vitalilty/Discovery program. The investigators plan to compare the effectiveness standard intervention (control) that includes text messaging aimed at encouraging cessation to four interventions: 1) choice of free (traditional) cessation aids (NRT: gum or patch), 2) free e-cigarettes, 3) Choice of free cessation aids (NRT or e-cigarettes) and reward based incentives for cessation, and 4) Choice of free cessation aids (NRT or e-cigarettes) and a virtual deposit-based incentives for cessation.

Primary outcome variable: Urine cotinine, anabasine, or blood carboxyhemoglobin testing (metabolites of nicotine) at 6 months following the quit date.

Secondary outcome variable: Urine cotinine, anabasine, or blood carboxyhemoglobin testing (metabolites of nicotine) at 1 month, 3 months, and 12 months following the quit date.

Background Tobacco use remains one of the most preventable causes of disease, disability, and death worldwide (CDC, 2014). Rates of smoking in the US have decreased to 18.1% in 2012 but remain far from the cessation goals set by tobacco prevention organizations (12% by 2020 in the US). To achieve these cessation goals and reduce harm from tobacco, the investigators need to both implement proven strategies to promote cessation and develop new approaches to increasing tobacco cessation (Frieden, 2014). Vitality is the wellness program for over 25 companies in the US. They are charged with providing a variety of wellness programs for the employees of companies they represent. These programs span a variety of health behaviors including tobacco use, obesity, healthy eating, driving while texting and many more.

Financial incentives have been effective in improving health in a variety of areas, including smoking cessation (Heil et al., 2008; Loewenstein et al., 2012; Lynagh et al., 2013; Sutherland et al., 2008; Volpp et al., 2009 ). In the largest (n = 878) and most successful trial, Volpp and colleagues (2009) found that financial incentives, totaling $750, increased long-term smoking cessation rates from 5.0% in the control group to 14.7% in the incentive group 12 months after quitting. Following a period of 6 months where incentives were discontinued this difference between groups remained intact, supporting the use of incentives for sustainable cessation efforts. Strong evidence supporting the use of incentives for smoking cessation and the allowance granted by the Affordable Care Act for employers to use up to 30% of total premiums for outcomes-based rewards or penalties has led to an increase in use of financial incentives by employers. An estimated 82% of large employers in 2013 used financial incentives to promote healthy behavior (Volpp, 2014). While financial incentives have been shown to improve rates of healthy behaviors, basic research in behavioral economics suggests that how you pay these incentives may be critical. Behavioral economics suggests that loss aversion may promote more behavior change than reward-based incentives. Whether or not this holds true in large employer based populations where participants are auto-enrolled has yet to be determined. The investigators propose conducting a 5- arm study examining the use of different financial incentive structures and new technologies to promote smoking cessation in Vitality members in the US. The relative effectiveness of how incentives are paid out is unknown. To shed light on this fundamental question the investigators will examine how incentives for assistance in quitting compare to incentives delivered for evidence of smoking abstinence and deposit contracts. Additionally the utility of e-cigarettes in promoting abstinence is not well understood. The use of e-cigarettes and other smoking cessation tools will be promoted and provided across all experimental arms so that the of the effectiveness of these aides can also be evaluated. The primary objective will be to identify differences in long-term abstinence rates. Secondary objectives include assessing sustained abstinence at follow-up. An opt-out enrollment procedure will be used for this study. All participants will have previously tested positive for cotinine and reported being a smoker, will be 18 years of age or older, will be a beneficiary of Vitality, and will have the opportunity to terminate their participation at any time. Employing an opt-out design for this trial will help to connect high-risk smokers, who are largely interested in changing their behavior, to potentially helpful treatments that they may not otherwise seek out. Below we describe the many reasons why an opt-out enrollment is appropriate for this trial. 1) An opt-out design is essential to answer the questions we are interested in: what rates of sustained smoking abstinence might an insurer expect to generate if it actually rolled out the interventions to be tested among its beneficiaries, and how do these interventions compare in terms of their effectiveness? Thus, in designing this trial, we explicitly aimed to mimic the roll out of a health initiative in a real-world setting; opt-out consent, whereby beneficiaries are engaged with the program unless they actively choose otherwise, is how such programs would be rolled out in the real world. As programs similar to the current trial are being developed and disseminated across the country it is imperative that we examine how interventions perform under these conditions. Enrolling large numbers of smokers in a study in which all will be offered some form of assistance with cessation provides high expected benefits, both to enrolled participants and in terms of the knowledge to be gained. While smoking rates have reduced to 18% in the United States, smoking related illness still remains the leading cause of preventable death in the United States. More than 75% of current American smokers wish to quit; 45% do quit for at least a day each year; and anti-smoking policies, new pharmaceuticals, and behavioral modification programs offer promise to help them. Nevertheless, only 2-3% of smokers attain prolonged abstinence annually. Given this high interest in quitting smoking, and low rates of successfully sustaining quit attempts with currently available programs, opt-out consent will ensure that all smokers will have the same access to potentially helpful programs without the added barrier of completing a lengthy enrollment/consent process. Vitality is committed to using the most effective means of reducing major risks to health in its membership and employee base. In order to achieve this goal they are working with innovative researchers at the University of Pennsylvania Center for Health Incentives and Behavioral Economics (CHIBE). Within the Vitality US population 13% of members tested positive for tobacco use. In the South African Vitality employee population smoking prevalence is estimated at 22%. Vitality is launching a study on tobacco cessation using incentives and new nicotine technologies for members in the US. Findings of the study will be published and used for development of a smoking cessation program offerings for Vitality. If successful this trial could serve as a model for other organizations interested in implementing a similar program. This study will use the National Institute on Aging supported Way to Health technology (RC2-AG036592) which has been used in many previous studies of this nature. As outlined in the Appendix, this web-based behavioral research infrastructure will substantially increase the efficiency of patient enrollment and tracking, data management, and incentive collection and disbursement, thereby enabling much larger studies than was possible previously.

Participants eligible for this trial will have been previously identified by the Vitality/Discovery group during various assessments they have conducted. All who meet our minimum eligibility requirements (18 years or older, smoke at least 5 cigarettes a day, tested positive for cotinine at a previous health screening) will be automatically enrolled into this study and randomized to one of four experimental arms and a control arm. All participants will be enrolled on the same day. Furthermore, all participants will be given the same quit date, a date one month from enrollment. This program will require participants to indicate their smoking status and provide samples for verification of abstinence at pre-determined dates after their quit date (1 month, 3 months, 6 months and 12 months post quit date). Participants who report having successfully quit will be asked to undergo a urine cotinine and anabasine test at 1 month, 3 months,6 months, and 12 months following their quit date. Cotinine will be used to determine abstinence in participants not reporting the use of NRT or ecigarettes. Anabasine will be used to determine abstinence for participants reporting use of NRT or ecigarettes, as cotinine tests cannot distinguish cigarette nicotine from replacement therapy nicotine. Participants who test positive for both cotinine and anabasine but report using only e-cigarettes and no other tobacco products will be asked to submit to a secondary test to determine abstinence. This test will be a blood carboxyhemoglobin test. Control Arm: Participants randomized to this arm will receive a standardized Vitality program aimed at promoting tobacco cessation. This program includes existing employee benefits for quitting and the use of text/email messages to encourage tobacco cessation. No incentives will be given to participants randomized to this arm. Free cessation aids will not be available to participants in this arm. They will receive compensation for completing study related activities (sample submissions). E-cigarette arm (Arm 2): Participants randomized to this experimental arm will receive the standardized program including text/email messaging and will have access to free e-cigarettes only. These products can be ordered directly, free of charge, through the web-based interface. No incentives will be given to participants randomized to this arm. They will receive compensation for completing study related activities (sample submissions). E-cigarette/NRT/Zyban/Chantix Choice arm (Arm 3): Participants randomized to this experimental arm will receive the standardized program including text/email messaging and will have access to free e-cigarettes, conventional Nicotine Replacement Therapy (NRT), Zyban, or Chantix. Each of these can be ordered directly, free of charge, through the web-based interface. No incentives will be given to participants randomized to this arm. They will receive compensation for completing study related activities (sample submissions). Outcome Incentive arm (Arm 4): Participants randomized to this experimental arm will receive the standardized program and access to free e-cigarettes, NRT, Zyban, or Chantix. In addition, they will also be able to earn incentives across six months for testing negative for tobacco use (see Incentive payout, below). They will also receive compensation for completing study related activities (sample submissions). Loss framing incentive arm (Arm 5): Participants randomized to this experimental arm will receive the standardized program and access to free e-cigarettes, NRT, Zyban, or Chantix. In addition they will also be able to earn incentives across six months through a pre-funded deposit or precommitment account. They will be notified that an incentive has been placed into an account for them. At each time point they will lose a portion of this initial funding if they do not provide biochemical evidence of abstinence. They will also receive compensation for completing study related activities (sample submissions).

ELIGIBILITY:
Inclusion Criteria:

* Vitality beneficiary
* 18 years or older
* reported and/or tested positive for being a smoker
* all participants will be able to opt-out of this program.

Exclusion Criteria:

* Participants who express wanting to opt-out of this program will be un-enrolled and excluded

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6006 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2016-11-05 (Actual); Study Completion 2017-04-20 (Actual)

PRIMARY OUTCOMES:
verified abstinence 6 months | 6 months
  Biometric testing (metabolites of nicotine) at 6 months following the quit date

SECONDARY OUTCOMES:
verified abstinence 1 months | 12 months
  Biometric testing (metabolites of nicotine) at 1 month, 3 months, and 12 months following the quit date.
verified abstinence 3 months | 12 months
  Biometric testing (metabolites of nicotine) at 1 month, 3 months, and 12 months following the quit date.
verified abstinence 12 months | 12 months
  Biometric testing (metabolites of nicotine) at 1 month, 3 months, and 12 months following the quit date.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Harhay MO, Troxel AB, Brophy C, Saulsgiver K, Volpp KG, Halpern SD. Financial Incentives Promote Smoking Cessation Directly, Not by Increasing Use of Cessation Aids. Ann Am Thorac Soc. 2019 Feb;16(2):280-282. doi: 10.1513/AnnalsATS.201808-574RL. No abstract available. PMID 30290121
- [Derived] Halpern SD, Harhay MO, Saulsgiver K, Brophy C, Troxel AB, Volpp KG. A Pragmatic Trial of E-Cigarettes, Incentives, and Drugs for Smoking Cessation. N Engl J Med. 2018 Jun 14;378(24):2302-2310. doi: 10.1056/NEJMsa1715757. Epub 2018 May 23. PMID 29791259